CLINICAL TRIAL: NCT05837351
Title: The CARE Project: Collaborative Adolescent Running Experience
Brief Title: The CARE (Collaborative Adolescent Running Experience) Project
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Richard Dopp, Associate Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00212052
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Depression; Anxiety; Major Depressive Disorder; Bipolar Disorder
Keywords: Running; Adolescents
MeSH Terms: conditions — Depression; Anxiety Disorders; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise -Running (Experimental)
  Interventions: Behavioral: Exercise -Running

INTERVENTIONS:
Behavioral: Exercise -Running — At baseline participants will wear a Fitbit for one week and attend the Runner's Assessment. After this the participant will begin to run 3 times per week for eight weeks. Every week, participation in a virtual support group with the physical therapist, research coordinator, and other research staff will be expected. Rest-activity cycles' data will be monitored; if at any point the runner is not able to complete 3 runs per week, participants will be encouraged to contact research staff the issues for this (such as medical problem or scheduling difficulty) and formulate plans to remediate the situation. Participants that would like to continue the treatment for an additional eight weeks will have additional data collected.
  Participants will also wear the Fitbit through-out the study and complete surveys during the study and have blood drawn.

SUMMARY:
This study is being completed to see if participants activity levels may have an impact as a treatment for depression, or depressive symptoms.

Eligible participants will be enrolled and have an 8-week running intervention three times each week.

The study hypothesizes that adolescents with Psychiatric disorders that are experiencing depressive symptoms will participate in a supported running intervention.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric disorders that are experiencing depressive symptoms (defined by the protocol)
* Must have a smart phone
* Parents/guardians will be advised to discuss their child's participation in the intervention with the participant's primary care physician

Exclusion Criteria:

* Adolescents with unstable cardiac, pulmonary, endocrine or renal disorders
* Adolescents with previous injuries or other conditions that may impact the safety of a running intervention

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The number of completed running sessions | weeks 1-8 during treatment period
  Feasibility and acceptability of the study will be the completion of running sessions based on the Fitbit and or self-report.

SECONDARY OUTCOMES:
Change in depression severity as reported by The Patient Health Questionnaire for Adolescents (PHQ-A) | Baseline (prior to treatment), 8 weeks (post intervention)
  This is a self-report questionnaire designed for the purpose of assessing anxiety, mood, eating, and substance use disorders. For the first section (9 questions) the participants will select from Not at all (0) to nearly every day (3).
  The next section asks if in the past year participants felt depressed or sad most days (yes or no) and if so, not difficult at all to extremely difficult. The last question participants are asked about suicide. Scores of 5, 10, 15, and 20 represent cut points for mild, moderate, moderately severe and severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dopp, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No